CLINICAL TRIAL: NCT07016620
Title: In-Office Transperineal Laser Ablation (TPLA) as a Salvage Treatment for Obstructive Benign Prostatic Hyperplasia (BPH) After Minimally Invasive Surgical Therapies (MIST)
Brief Title: Laser Ablation a Salvage Treatment for Obstructive Benign Prostatic Hyperplasia
Acronym: ECHOLASER
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Rocamed Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: 25-327
Record Dates: First submitted 2025-04-08; First posted 2025-06-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: benign prostatic hyperplasia (BPH); lower urinary tract symptoms (LUTS); transperineal Laser Ablation (TPLA); Minimally Invasive Surgical Therapies (MIST); salvage treatment
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transperineal Laser Ablation (TPLA): Patients with recurrent Benign Prostatic Hyperplasia (BPH) after Minimally Invasive Surgical Therapies previous (MIST)
  Interventions: Procedure: Transperineal Laser Ablation (TPLA)

INTERVENTIONS:
Procedure: Transperineal Laser Ablation (TPLA) — Outpatient treatment with Transperineal Laser Ablation (TPLA) as a salvage therapy after previous Minimally Invasive Surgical Therapies (MIST)

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common condition affecting aging men, often leading to lower urinary tract symptoms (LUTS). While Minimally Invasive Surgical Therapies (MIST) procedures offer less invasive alternatives to traditional surgery, some patients experience symptom recurrence or require further intervention due to lack of adequate relief of obstruction. Treatment of persistent obstruction after MIST therapy (BPH salvage therapy) typically requires surgical intervention like transurethral resection of prostate (TURP). This study proposes to evaluate the effectiveness of in-office transperineal laser ablation (TPLA) using the Echolaser system as a minimally invasive treatment option for these patients, potentially avoiding more invasive surgical procedures. The Cleveland Clinic sees a high volume of BPH salvage patients, making this an ideal setting for this research.

DETAILED DESCRIPTION:
TPLA of the prostate represents a promising minimally invasive treatment modality for men experiencing LUTS secondary to BPH. This technique offers a potentially attractive alternative to traditional surgical interventions, particularly given the growing interest in less invasive procedures. The current literature focuses on evaluating the effectiveness of TPLA in improving urodynamic parameters (specifically maximum urinary flow rate (Qmax) and post-void residual volume (PVR), alleviating LUTS, and preserving sexual and ejaculatory function, as well as surgical complications.

In a recent systematic review, which included 6 studies, studies consistently reported statistically significant improvements from baseline in Qmax, PVR, and IPSS scores (International Prostate Symptom Score) at all measured time points. Furthermore, three of the studies demonstrated that TPLA did not negatively impact sexual function, showing no significant changes in IIEF-6 scores (International Index of Erectile Function) and, in some cases, statistically significant improvements in MSHQ-EjD scores (Male Sexual Health Questionnaire) at various follow-up intervals, Low complication rates were observed across all studies. Pooled analysis of the available data revealed clinically meaningful improvements in both voiding and sexual function outcomes at 1-, 3-, and 6-, and 12-months post-treatment, when compared to baseline values.

While the preliminary findings from these pilot studies suggest that TPLA may be a valuable treatment option for BPH, further research is warranted. Specifically, there is a lack of data demonstrating the efficacy of TPLA as a salvage option, where other MIST options failed.

ELIGIBILITY:
Inclusion Criteria:

* Men > 40 years old
* History of Minimally invasive BPH procedure within the last 5 years.
* IPSS >= 12
* Prostate Volume 30 - 80 gr as assessed by CT, MRI or TRUS.
* PSA <4 or for patients with PSA 4-10 evaluation has been performed to rule out prostate cancer using biopsy, MRI, biomarker, or surgeon judgement. Labs within 1 year of study initiation
* PVR > 150cc or reduced flow on uroflow likely due to obstruction based on clinical judgement
* IIEF-6>or =10 without medication

Exclusion Criteria:

* Indwelling catheter or intermittent catheterization
* History of urethral strictures
* Previous diagnosis of Prostate cancer
* Active UTI or prostatitis
* Hypoactive detrusor function
* Neurogenic bladder (secondary to stroke, Multiple Sclerosis, Parkinson's disease, Spinal cord injury)
* Ejaculatory dysfunction (retrograde ejaculation, anorgasmia or anejaculation)
* Prior traditional BPH surgery (TURP, PVP, Aquablation, HOLEP, SP)
* Presence of obstructive median lobe
* Moderate to severe or severe ED based on IIEF-6/SHIM (SHIM of 10)
* Peyronie's disease

Min Age: 40 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Benign Prostatic Hyperplasia (BPH) only occurs in men
Study Population: Benign Prostatic Hyperplasia (BPH) salvage therapy patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of in-office TPLA on voiding function in patients with recurrent BPH after prior MIST procedures | baseline, and then 1-, 3-, 6- and 12-months post-treatment with laser ablation
  Change in Urinary Function as measured with IPSS score, Uroflow variables (Qmax) and Post void residue (PVR)

SECONDARY OUTCOMES:
Evaluate the effect of TPLA on erectile function & ejaculatory functions in this patient population | baseline, and then 1-, 3-, 6- and 12-months post-treatment with laser ablation
  Change in Sexual function as measured by IIEF 6, MSHQ-EjD

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sessa F, Bisegna C, Polverino P, Gacci M, Siena G, Cocci A, Li Marzi V, Minervini A, Serni S, Campi R. Transperineal laser ablation of the prostate (TPLA) for selected patients with lower urinary tract symptoms due to benign prostatic obstruction: a step-by-step guide. Urol Video J. 2022;15:100167. doi:10.1016/j.urolvj.2022.100167.
- [Result] Tafuri A, Panunzio A, De Carlo F, Luperto E, Di Cosmo F, Cavaliere A, Rizzo M, Tian Z, Shakir A, De Mitri R, Porcaro AB, Cerruto MA, Antonelli A, Cormio L, Carrieri G, Karakiewicz PI, Abreu AL, Pagliarulo V. Transperineal Laser Ablation for Benign Prostatic Enlargement: A Systematic Review and Pooled Analysis of Pilot Studies. J Clin Med. 2023 Feb 26;12(5):1860. doi: 10.3390/jcm12051860. PMID 36902647
- [Result] de Rienzo G, Lorusso A, Minafra P, Zingarelli M, Papapicco G, Lucarelli G, Battaglia M, Ditonno P. Transperineal interstitial laser ablation of the prostate, a novel option for minimally invasive treatment of benign prostatic obstruction. Eur Urol. 2021 Jul;80(1):95-103. doi: 10.1016/j.eururo.2020.08.018. Epub 2020 Aug 28. PMID 32868137
- [Result] Manenti G, Perretta T, Calcagni A, Ferrari D, Ryan CP, Fraioli F, Meucci R, Malizia A, Iacovelli V, Agro EF, Floris R. 3-T MRI and clinical validation of ultrasound-guided transperineal laser ablation of benign prostatic hyperplasia. Eur Radiol Exp. 2021 Sep 17;5(1):41. doi: 10.1186/s41747-021-00239-9. PMID 34532768